CLINICAL TRIAL: NCT05306847
Title: Sintilimab Combined With Anlotinib Therapy for Patients With Initially Unresectable Stage II-III Non-small Cell Lung Cancer: A Prospective, Single-arm Study
Brief Title: Sintilimab Combined With Anlotinib Therapy for Initially Unresectable Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Xinda Biopharmaceutical Group (Unknown); Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, YueJuan Cheng, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-3340
Record Dates: First submitted 2022-03-21; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small-cell lung cancer; Sintilimab; Anlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Sintilimab will be given intravenously at a dose of 200mg every 21 days. Anlotinib will be given at a dose of 12mg once daily on days 1-14 of a 21-day cycle.
  Tumor evaluation will be conducted after treatment of the tested regimen every 2 cycles. Subsequent treatment will be determined based on the evaluation results: If the patients are not suitable for radical surgery, but the result of efficacy evaluation is CR, PR, or SD, they can continue to receive the tested regimen. If the patients are still not suitable for radical surgery after 6 cycles of the tested regimen, the standard first-line or immunotherapy after chemoradiotherapy or radiotherapy will be given. If patients are eligible for radical surgery, surgery will be performed within 4 weeks after completion of the last tested regimen.
  Interventions: Drug: Sintilimab; Drug: Anlotinib

INTERVENTIONS:
Drug: Sintilimab — Sintilimab will be given intravenously at a dose of 200mg every 21 days.
  Other Names: IBI308; Tyvyt
Drug: Anlotinib — Anlotinib will be given at a dose of 12mg once daily on days 1-14 of a 21-day cycle.
  Other Names: Anlotinib hydrochloride; AL3818

SUMMARY:
Concurrent or sequential chemoradiotherapy has been recommended as the standard treatment for locally advanced and unresectable non-small cell lung cancer (NSCLC). However, its efficacy remains to be improved. PD-1/PD-L1 inhibitors have been proven to be effective for late-stage NSCLC, and anti-angiogenesis agents have also been used for the first-line treatment of advanced or metastatic NSCLC. Therefore, we designed this single-arm clinical trial, which aims to investigate the safety and feasibility of sintilimab combined with anlotinib therapy for patients with initially unresectable stage II-III NSCLC.

DETAILED DESCRIPTION:
Concurrent or sequential chemoradiotherapy is the standard treatment for patients with locally advanced NSCLC, but patients receiving chemoradiotherapy have limited improvement in prognosis and are almost impossible to achieve a radical cure. Considering the excellent effect of immunotherapy and anti-angiogenesis therapy in NSCLC, we designed this single-arm clinical study, which aims to investigate the safety and feasibility of sintilimab combined with anlotinib therapy for patients with initially unresectable stage II-III NSCLC, in order to enable patients to achieve further surgical treatment and prolonged survival.

ELIGIBILITY:
Inclusion Criteria:

1. According to the 8th edition of the AJCC/UICC TNM staging system for NSCLC, patients with locally advanced (stage II-III C) NSCLC confirmed by histology who are initially unable to undergo surgery and concomitant radiochemotherapy and are confirmed to have at least one measurable lesion according to RECIST 1.1.
2. Age ≥18 years and ≤75 years.
3. ECOG PS score: 0 to 1.
4. The main organs function is normal, that is, the following criteria met:

   1. Good hematopoietic function, defined as absolute neutrophil count ≥1.5×109 /L, platelet count≥100 ×109 /L, hemoglobin ≥90g/L [no blood transfusion or no erythropoietin (EPO) dependence within 7 days before enrollment];
   2. Biochemical test results should meet the following criteria: BIL < 1.25 times the upper limit of normal value (ULN); ALT and AST < 2.5 × ULN; in case of liver metastases, ALT and AST < 5 × ULN; Cr ≤1.5×ULN or creatinine clearance (CCr) ≥60ml/min; Coagulation function is good, INR and PT ≤1.5 × ULN;
   3. The oxygen saturation of the finger tip ≥ 92% both at rest and during walking (without oxygen inhalation).
5. The life expectancy ≥12 weeks.
6. Signed and dated informed consent.

Exclusion Criteria:

1. Subjects at risk of massive hemoptysis or with blood in sputum, including but not limited to tumor lesions no more than 5 mm away from large vessels, tumors invading large vessels, and obvious lung cavity/necrotizing tumors.
2. Small cell lung cancer (including mixed small cell and non-small cell lung cancer) or central squamous cell carcinoma.
3. With driver mutation (EGFR/ALK/ROS1).
4. With uncontrollable hypertension (systolic pressure > 160 mmHg, diastolic pressure > 100 mmHg) even receiving antihypertensive drug therapy.
5. Has an active autoimmune disease, history of allogeneic stem cell transplantation or organ transplantation that has required systemic treatment. Replacement therapy is not considered a form of systemic treatment and is allowed.
6. Has an active infection requiring systemic therapy.
7. Has other malignant tumors (except radical cervical carcinoma in situ, non-melanoma skin cancer, etc.) or concomitant diseases that seriously endanger the patients or affect the patients completing the study at the same time.
8. With immunodeficiency status, including but not limited to HIV infection and primary immunodeficiency diseases.
9. Previously treated with ICIs.
10. Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Surgical conversion rate | 18 weeks from the initiation of the tested regime therapy
  The surgical conversion rate was defined as the proportion of subjects with the successful conversion over all subjects who received the tested regime.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 18 weeks from the initiation of the tested regime therapy
  ORR is defined as the percentage of participants who have the best overall response (BOR) of complete response (CR) or partial response (PR) assessed based on RECIST 1.1.
R0 resection rate | within 28 working days after operation
  R0 resection rate is defined as the complete resection rate of all tumor under microscope.
Major pathological response rate | within 28 working days after operation
  Major pathological response rate is defined as the percentage of patients who achieved a major pathological response (residual tumor ≤10%).
Pathological complete response rate | within 28 working days after operation
  Pathological complete response rate is defined as the percentage of patients who achieved a pathological complete response (residual tumor = 0%).
Overall survival (OS) | 2 years from the initiation of the tested regime therapy
  OS is measured from the time from the treatment onset (date of first study dose) until the date of death from any cause.
Progression-free survival (PFS) | 2 years from the initiation of the tested regime therapy
  PFS is measured from the time from the treatment onset (date of first study dose) until the date of tumor progression or death from any cause.
Disease-free survival (DFS) | 2 years from the initiation of the tested regime therapy
  DFS is measured from the time from radical surgery until the date of tumor progression or death from any cause.
Treatment-related adverse events | 3 months from the end of the tested regime therapy
  Incidence and grade of treatment-related adverse events assessed based on CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Chunmei Bai, Professor, Principal Investigator — Peking union medical colloge hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 1 year of study completion
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick S, Brahmer J, Swanson SJ et al: Nivolumab (NIVO) + platinum-doublet chemotherapy (chemo) vs chemo as neoadjuvant treatment (tx) for resectable (IB-IIIA) non-small cell lung cancer (NSCLC) in the phase 3 CheckMate 816 trial. Cancer research 2021, 81(13 SUPPL).
- [Background] Mery B, Guy JB, Swalduz A, Vallard A, Guibert C, Almokhles H, Ben Mrad M, Rivoirard R, Falk AT, Fournel P, Magne N. The evolving locally-advanced non-small cell lung cancer landscape: Building on past evidence and experience. Crit Rev Oncol Hematol. 2015 Nov;96(2):319-27. doi: 10.1016/j.critrevonc.2015.05.020. Epub 2015 Jun 7. PMID 26095618
- [Background] Faivre-Finn C, Vicente D, Kurata T, Planchard D, Paz-Ares L, Vansteenkiste JF, Spigel DR, Garassino MC, Reck M, Senan S, Naidoo J, Rimner A, Wu YL, Gray JE, Ozguroglu M, Lee KH, Cho BC, Kato T, de Wit M, Newton M, Wang L, Thiyagarajah P, Antonia SJ. Four-Year Survival With Durvalumab After Chemoradiotherapy in Stage III NSCLC-an Update From the PACIFIC Trial. J Thorac Oncol. 2021 May;16(5):860-867. doi: 10.1016/j.jtho.2020.12.015. Epub 2021 Jan 19. PMID 33476803
- [Background] De Ruysscher D, Botterweck A, Dirx M, Pijls-Johannesma M, Wanders R, Hochstenbag M, Dingemans AM, Bootsma G, Geraedts W, Simons J, Pitz C, Lambin P. Eligibility for concurrent chemotherapy and radiotherapy of locally advanced lung cancer patients: a prospective, population-based study. Ann Oncol. 2009 Jan;20(1):98-102. doi: 10.1093/annonc/mdn559. Epub 2008 Aug 20. PMID 18718891
- [Background] Xiao W, Hong M. Concurrent vs sequential chemoradiotherapy for patients with advanced non-small-cell lung cancer: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2021 Mar 19;100(11):e21455. doi: 10.1097/MD.0000000000021455. PMID 33725921
- [Background] Eberhardt WE, Pottgen C, Gauler TC, Friedel G, Veit S, Heinrich V, Welter S, Budach W, Spengler W, Kimmich M, Fischer B, Schmidberger H, De Ruysscher D, Belka C, Cordes S, Hepp R, Lutke-Brintrup D, Lehmann N, Schuler M, Jockel KH, Stamatis G, Stuschke M. Phase III Study of Surgery Versus Definitive Concurrent Chemoradiotherapy Boost in Patients With Resectable Stage IIIA(N2) and Selected IIIB Non-Small-Cell Lung Cancer After Induction Chemotherapy and Concurrent Chemoradiotherapy (ESPATUE). J Clin Oncol. 2015 Dec 10;33(35):4194-201. doi: 10.1200/JCO.2015.62.6812. Epub 2015 Nov 2. PMID 26527789
- [Background] Deng H, Liu J, Cai X, Chen J, Rocco G, Petersen RH, Brunelli A, Ng CSH, D'Amico TA, Liang W, He J. Radical Minimally Invasive Surgery After Immuno-chemotherapy in Initially-unresectable Stage IIIB Non-small cell Lung Cancer. Ann Surg. 2022 Mar 1;275(3):e600-e602. doi: 10.1097/SLA.0000000000005233. PMID 34596079
- [Background] Chu T, Zhong R, Zhong H, Zhang B, Zhang W, Shi C, Qian J, Zhang Y, Chang Q, Zhang X, Dong Y, Teng J, Gao Z, Qiang H, Nie W, Zhao Y, Han Y, Chen Y, Han B. Phase 1b Study of Sintilimab Plus Anlotinib as First-line Therapy in Patients With Advanced NSCLC. J Thorac Oncol. 2021 Apr;16(4):643-652. doi: 10.1016/j.jtho.2020.11.026. Epub 2021 Jan 29. PMID 33524601